CLINICAL TRIAL: NCT04717648
Title: The Effect of Postoperative C-Reactive Protein and Sodium Value on the Early Prediction of Anastomotic Leaks in Patients Operated on for Colorectal Cancer
Brief Title: C-Reactive Protein and Sodium in Predicting Anastomotic Leakage
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semra Demirli Atici, Principal Investigator, Tepecik Training and Research Hospital
Other Study IDs: 2020/13-51
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer
Keywords: anastomotic leak; hyponatremia; colorectal carcinoma; c-reactive protein
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak; Hyponatremia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with anastomotic leakage: Post operative anastomotic leakage
  Interventions: Diagnostic Test: Biochemical test
- Patients without anastomotic leakage: Post operative without anastomotic leakage
  Interventions: Diagnostic Test: Biochemical test

INTERVENTIONS:
Diagnostic Test: Biochemical test — C Reactive protein and sodium

SUMMARY:
Anastomotic leakage is serious morbidity that can develop in patients operated on for colorectal cancer and can reach potentially life-threatening dimensions. Many international studies have been conducted to reduce and eliminate this postoperative complication that may have a mortal course. In these studies, preoperative, perioperative and postoperative factors of the patient, operation techniques, structure of the material used in the operation and multiple factors belonging to the surgeon were held responsible. Intraabdominal sepsis secondary to late anastomotic leakage and subsequent multiorgan failure can cost the patient's life. Anastomotic leaks that develop in patients who have been operated for colorectal cancer; In order to detect patients' postoperative clinical findings, laboratory examinations, imaging tests, and to eliminate them before intraabdominal sepsis develops, studies including many different laboratory and imaging methods have been carried out. Although previous studies have shown that there are many laboratory examinations and imaging methods that can predict anastomotic leaks early, they have many advantages over each other in terms of efficiency, sensitivity, specificity, and cost.

The investigators aimed to investigate the effectiveness of C reactive protein and blood sodium value, as well as their superiority, among the tests that can predict postoperative anastomotic leakage, especially in patients who have undergone a single anastomosis following resection for non-metastatic colorectal cancer.

DETAILED DESCRIPTION:
* Investigate the effectiveness of postoperative C-reactive protein and sodium values in predicting anastomotic leakage in the early postoperative period in patients who have undergone anastomosis following resection for non-metastatic colorectal cancer, and their superiority to each other.
* Investigate the effectiveness of these laboratory parameters in developing anastomotic leaks according to tumor location and different age subgroups (<45 years, 45-65 years,> 65 years).

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 who were operated due to elective colorectal cancer
2. Patients who are known to have no solid organ metastases in preoperative imaging methods and whose perioperative surgery notes support this finding
3. Patients with ileocolic, colocolic, colorectal anastomosis during the operation
4. Patients whose postoperative 1,3,5th day C- Reactive protein and sodium values were measured

Exclusion Criteria:

1. Patients under the age of 18
2. Emergency operated patients
3. Patients on a routine dialysis program due to Chronic renal failure
4. Patients with a known diagnosis of liver cirrhosis
5. Patients who are irresectable during the operation and therefore have undergone palliative surgery
6. Patients whose C- Reactive protein and Sodium values were not measured on the postoperative 1, 3, 5th day
7. Patients with abdominoperineal resection and no bowel anastomosis during the operation
8. Patients who have not undergone ileocolic, colocolic, colorectal or ileorectal anastomosis during the operation.
9. Patients found to be metastatic during the operation
10. Patients who have undergone additional surgical resection (metastasectomy, etc.) due to solid organ metastasis during the operation
11. Patients who have had more than one gastrointestinal anastomosis during the same surgery
12. Patients undergoing concurrent hyperthermic intraperitoneal chemotherapy (HIPEC) and / or cytoreductive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Early predictive factors of anastomotic leakege | 2 or 3 days
  The anastomotic leak of the measurement The measurement tool is the laboratory parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided